CLINICAL TRIAL: NCT07163780
Title: The Effectiveness of the HEP (Homeostasis-Enrichment-Plasticity) Approach in Infants With Down Syndrome
Brief Title: The Effect of the HEP Approach in Infants With Down Syndrome
Acronym: HEP-DS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izgi Miray Demirbag (Other)
Responsible Party: Sponsor-Investigator, Izgi Miray Demirbag, Physiotherapist, Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-10840098-202.3.02-2211
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Down Syndrome (DS)
Keywords: Down Syndrome; Infants; Early Intervention; Neuroplasticity; Environmental Enrichment
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: The study includes two groups: one group will receive the HEP intervention, and the other group will receive traditional therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEP Intervention (Experimental): Participants will receive 12 sessions of HEP therapy, once per week, 45 minutes each.
  Interventions: Behavioral: HEP Intervention
- Traditional Therapy (Active Comparator): Participants will receive 12 sessions of traditional therapy, once per week, 45 minutes each.
  Interventions: Behavioral: Traditional Therapy

INTERVENTIONS:
Behavioral: HEP Intervention — This intervention is administered to the HEP Intervention arm.
  The HEP approach, which includes intervention, is a child-centered, family-based early intervention approach based on the principles of enriched environment and plasticity, emphasizing the importance of homeostasis. It is based on theories that argue that development occurs as a result of the dynamic interaction between the environment, time, task, and individual (Ecological Theory, Dynamic Systems Theory, Perception-Action Theory, Neuronal Group Selection Theory, and the Person-Environment-Occupation Model). Hypotheses for intervention are generated based on a comprehensive assessment of these four fundamental factors (environment, time, task, and individual), and 10 core principles derived from environmental enrichment studies are applied with the guidance of ecological models.
  Arms: HEP Intervention
Behavioral: Traditional Therapy — Participants in this arm will receive conventional pediatric therapy, consisting of 12 weekly sessions of 45 minutes each. Sessions will focus on standard motor and sensory development exercises, delivered by a physical therapist experienced in pediatric rehabilitation.
  Arms: Traditional Therapy

SUMMARY:
This study evaluates the effect of the HEP (Homeostasis-Enrichment-Plasticity) approach on motor and sensory development in infants with Down syndrome. Thirty-two infants will receive either HEP or traditional therapy over 12 sessions, and outcomes will be measured using standardized developmental tests.

DETAILED DESCRIPTION:
This clinical study will be conducted at a private clinic in Istanbul and will enroll 26 infants with Down syndrome who meet the inclusion criteria. Participants will be recruited through social media and referrals from professionals who follow infants with Down syndrome.

Written informed consent will be obtained from parents after explaining the study's purpose, duration, assessments, and interventions. Demographic, perinatal, natal, and postnatal data will be collected via a "Demographic Information Form." Gross and fine motor skills will be evaluated with Peabody Developmental Motor Scales-2 (PDMS-2), sensory functions with the Infant Sensory Function Test (BDFT), and parents will complete the The Ages and Stages Questionnaires (ASQ) to assess multiple developmental domains. Individual goals will be set using the Goal Attainment Scale (GAS), and social validity will be assessed post-intervention via a parent questionnaire.

The intervention group will receive 12 sessions (once a week, 45 minutes each) of HEP therapy, delivered by a physiotherapist experienced in the HEP approach. The control group will receive 12 sessions of traditional therapy administered by an experienced pediatric rehabilitation physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 4 and 12 months old
* Must have been diagnosed with Down Syndrome
* Must not be at any neurological risk
* Parent must agree to participate regularly in the study process

Exclusion Criteria:

* History of intraventricular hemorrhage (Grade III or IV)
* Major vision or hearing impairment
* History of febrile convulsion
* Medical conditions (e.g., oxygen dependence) that prevent active participation in the study
* Participation in other experimental rehabilitation studies

Ages: 4 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2025-12-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scales-2 (PDMS-2) | Pre-intervention and 12-week post-intervention.
  The PDMS-2 is a scale used to identify motor developmental delays in children aged 0-6 and to determine motor skill levels and individual needs.
  The PDMS-2 consists of two main sections: gross motor and fine motor, and 249 items. The gross motor section consists of reflexes, balance, locomotion, and object manipulation, while the fine motor section consists of comprehension and visual-motor integration. A score of 2 is given if the child's performance is within the desired level, 1 if it is similar to the desired level, and 0 if it is not.
  To determine the risk and level of developmental delay, gross motor skills, fine motor skills, and general motor development are categorized as "very low, low, below average, average, above average, high, and very high," using age-appropriate normative ranges in the test manual.

SECONDARY OUTCOMES:
Test of Sensory Functions in Infants (TSFI) | Pre-intervention and 12-week post-intervention.
  Developed to assess sensory responsiveness, this test consists of five subsections and 24 items, and takes 20 minutes to administer. The test subsections include tactile deep pressure response, adaptive motor functions, visual-tactile integration, oculomotor control, and vestibular stimulus response.
  This test is suitable for evaluating at-risk groups for sensory processing disorders, such as infants with developmental delays. Based on their score, the infant is assessed as normal, at-risk, or impaired in terms of sensory processing. A higher score indicates better sensory processing.
The Ages and Stages Questionnaires (ASQ) | Pre-intervention and 12-week post-intervention.
  The ASQ is a developmental screening test that allows parents to assess a child's development. The questionnaires consist of three sections: demographic questions, a 30-question section about the child's development, and seven open-ended questions. The 30 questions addressing the child's development cover the areas of communication, fine motor development, gross motor development, problem-solving, and personal and social development, with each section consisting of six questions.

OTHER OUTCOMES:
The Goal Attainment Scale (GAS) | Pre-intervention and 12-week post-intervention.
  The Goal Attainment Scale (GAS) is the most commonly recommended goal-setting methodology for measuring change during and after intervention in clinical and research applications. The GAS, which assesses the child's achievement of individual goals established with parents at the beginning of the intervention, is a reliable tool for children with developmental challenges and provides subjective information about the child's needs.
  The GAS has a rating scale of "-2" to "+2."

CONTACTS AND LOCATIONS:
Overall Officials: Aymen Balıkcı, Dr. Physiotherapist, Study Director
Locations (1):
- Sense On, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participant consent does not include sharing data with other researchers. Data will be maintained in strict confidentiality.